CLINICAL TRIAL: NCT03304067
Title: Digital Health Tool for Parental Management of Childhood Asthma -- Impact on Asthma Control Test Scores
Brief Title: Asthma Control Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evidation Health (Industry)
Collaborators: Tueo Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EH-005
Record Dates: First submitted 2017-10-02; First posted 2017-10-06 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Childhood Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Tueo Program
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Tueo Program — The asthma management solution utilizes devices (2 to attach on the child's bed and 1 for data transmission), which collect various metrics for a tailored smartphone application experience. The smartphone application provides access to view metrics from the devices, educational and clinical context content, and an asthma coach.
  Arms: Intervention

SUMMARY:
The "Digital Health Tool for Parental Management of Childhood Asthma -- Impact on Asthma Control Test Scores" Study is a 16 week, prospective, intent-to-treat, 2-arm randomized controlled trial that aims to evaluate the impact of the Tueo Health program on asthma control as indicated by change in baseline and study end (week 16) score on the Childhood Asthma Control Test score (ages 6- under 12 years) and the Asthma Control Test (ages 12-17 years) in children with uncontrolled asthma as the primary study objective.

ELIGIBILITY:
Inclusion Criteria:

* Parent has a child who is > 6 and < 17.5 years old
* Parent reports child has a diagnosis of asthma
* Child takes daily asthma controller medication
* Child has used rescue inhaler (e.g.albuterol, ProAir, etc) or nebulizer at least 2 times per week in the past 4 weeks
* Child sleeps on a toddler, single, or double bed by themselves
* Child will live in the same home for the majority of the next 16 weeks
* Parent is > 18 years old

Exclusion Criteria:

* Child's asthma has been controlled over the past 4 weeks
* Child has any of the following conditions: sleep apnea, congenital heart disease, cardiac arrhythmias, or any other heart abnormalities, neurologic conditions including seizures, cerebral palsy, muscular dystrophy, genetic conditions or developmental disorders, autism, other major medical condition
* Child is currently pregnant
* Child was born premature (earlier than 36 weeks)
* Parent is not fluent in English
* No in-home WiFi
* Parent does not use an Android phone as their primary phone
* In a household with an existing enrolled participant in the study, even for a different child (e.g. only one child in a household may have questions reported back to the researchers by their parent)
* Lives in Hawaii or Alaska

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Change in ACT/C-ACT scores | Baseline and Week 16
  Change in ACT/C-ACT scores from baseline to study end

CONTACTS AND LOCATIONS:
Locations (1):
- Evidation Health, San Mateo, California, United States

IPD SHARING:
Plan to Share IPD: No